CLINICAL TRIAL: NCT00485823
Title: The Assessment of a Weight Management Program for Treatment-Emergent Weight Gain in Patients With Schizophrenia, Schizophreniform Disorder, and Schizoaffective Disorder During Olanzapine Therapy
Brief Title: Assessment of a Weight Management Program for Weight Gain in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6696; F1D-KL-S031
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenic Disorders
MeSH Terms: conditions — Schizophrenia | interventions — olanzapine-fluoxetine combination

INTERVENTIONS:
Drug: Olanzapine Hydrochloride
Procedure: Weight Management Program

SUMMARY:
The purpose of this study is to develop the weight management program, which is combined with healthy diet, proper physical exercise, and behavior modification, related to patient's quality of life. The patients groups are in routine practice with 5-20 mg olanzapine. The study results may be utilized for patients who have gained weight on olanzapine and also other antipsychotic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 65 years (inclusive)
* Subjects must meet the DSM-IV criteria for schizophrenia, schizoaffective disorder, or schizophreniform disorder
* Subjects must have been treated with olanzapine (5 to 20 mg/day) for at least 12 weeks prior to study entry and who experienced a weight gain of greater than or equal to 7% of body weight during olanzapine treatment

Exclusion Criteria:

* Treatment with an injectable depot neuroleptic 14 days before visit 1
* Subjects with an PANSS score greater than 70
* One or more seizures without a clear and unresolved etiology
* Known diagnosis of DSM-IV substance dependence (except nicotine and caffeine) within the past 2 months, which in the opinion of the investigator is affecting the diet and/or weight of the subject
* As a result of liver function test, ALT/AST ranges are shown twice the upper limit of the normal reference range

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-12; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Comparison in the change in body weight from baseline to endpoint in the intervention group versus the control group

SECONDARY OUTCOMES:
Mean change from baseline to endpoint in the Stunkard and Messick Eating Inventory
Measure safety parameters, including medical history, psychiatric and physical examinations, vital signs (blood pressure, pulse and weight), clinical laboratory tests and record of symptoms
Severity of psychiatric symptoms and extrapyramidal symptoms were monitored using the PANSS and the AIMS, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com